CLINICAL TRIAL: NCT03435926
Title: Evaluating the Link Between Active Neovascularization Found on OCT and Eye Fixation Quality Measured With Microperimetry in ARMD Patients Treated With antiVEGF
Brief Title: OCT and Microperimetry in Patients With Active Neovascular ARMD (CORFI)
Acronym: CORFI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: I16021 (CORFI)
Record Dates: First submitted 2018-02-07; First posted 2018-02-19 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2018-09

CONDITIONS: Choroidal Neovascularization, Visual Field, Visual Acuity
MeSH Terms: conditions — Choroidal Neovascularization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
ARMD is the main cause of visual disability after 50 years old in France. Patients with active neovascular ARMD are treated with intravitreal injections of antiVEGF. Reinjections criteria are decrease of best corrected visual acuity or active neovascularization's signs (mostly found on macular OCT but also on angiography when necessary).

The aim of this study is to evaluate the link between active neovascularization found on OCT and eye fixation quality measured with microperimetry in ARMD patients treated with antiVEGF.

Quality of eye fixation and exudative signs presents or not present on OCT will be gathered at each consultation over the two-years follow-up for each patient. The mean central retinal sensitivity, the best corrected visual acuity and the bivariate contour ellipse area will also be gathered.

In case no link will be found, for instance bad fixation quality without exudative signs on OCT or good fixation stability despite exudative signs on OCT, microperimetry should have an interest to improve reinjections criteria with a treatment more suitable to the patient.

ELIGIBILITY:
Inclusion Criteria:

* patients > 50 years old,
* With neovascular ARMD
* who need an induction treatment (de novo patients or patients who had their last intravitreal injection of antiVEGF more than 6 months ago)

Exclusion Criteria:

* Other maculopathies
* Severe glaucoma with central visual field defect
* Diabetic patients
* Corneal, lens or vitreous opacities interfering in OCT analysis
* Attention or comprehension deficit

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with active neovascular ARMD treated with antiVEGF
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2018-02-13 (Actual); Primary Completion 2021-02-13 (Estimated); Study Completion 2021-02-13 (Estimated)

PRIMARY OUTCOMES:
fixation stability measured by microperimetry and exudative signs on OCT | 2 years
  quality of eye fixation and exudative signs presents or not present on OCT will be gathered at each consultation over the two-years follow-up.
  The fixation stability is classified as follows:
  * Stable if more than 75% of the fixation points are contained inside the circle of 2 degrees of diameter
  * Relatively unstable if more than 75% of the fixation points are contained within the circle of 4 degrees of diameter and less than 75% contained within that of 2 degrees of diameter
  * Unstable if less than 75% of the fixation points are contained within the circle of 4 degrees of diameter

SECONDARY OUTCOMES:
Bivariate Contour Ellipse Area (BCEA) value | 2 years
  BCEA will be gathered at each consultation over the two-years follow-up
mean central retinal sensitivity | 2 years
  mean central retinal sensitivity will be gathered at each consultation over the two-years follow-up
Best Corrected Visual Acuity (BCVA) | 2 years
  BCVA will be gathered at each consultation over the two-years follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Limoges, France

IPD SHARING:
Plan to Share IPD: No